CLINICAL TRIAL: NCT00192725
Title: Tryptophan Depletion in Acute Mania - A Randomized Controlled Trial
Brief Title: Tryptophan Depletion in Acute Mania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Beersheva Mental Health Center (Other Government)
Responsible Party: Ehud Klein, MD, Head Department of Psychiatry, Rambam Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tryp.dep.maniaCTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2005-09

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; acute mania; tryptophan depletion; placebo controlled add-on; Bipolar disorder- manic type
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

INTERVENTIONS:
Other: rapid tryptophan depletion — Amino-acid mixture without tryptophan

SUMMARY:
Serotonin (5-HT) is important in mood regulation and is believed to play a major role in the pathophysiology of major depression (MD). Selective serotonin reuptake inhibitors (SSRIs) are currently the most widely used drugs for the treatment of depression. Patients with bipolar disorder (BD) who are treated for depression with SSRIs might develop mania, which is believed to be triggered by antidepressant treatment. Rapid tryptophan depletion (RTD) has been shown to induce transient depressive symptoms in remitted depressed patients treated with SSRIs. In remitted manic patients treated with lithium, RTD does not seem to have clinical effects. However, RTD was not studied in acutely manic patients and could theoretically have antimanic properties. In this double blind randomized placebo controlled study RTD will be used as a tool to assess the role of 5-HT in mania and will be evaluated for its antimanic properties and potential use as augmentation to drug treatment in acute mania.

ELIGIBILITY:
Inclusion Criteria:

* Acute mania
* Ability to provide written informed consent

Exclusion Criteria:

* Mixed affective states
* Suicidal ideation
* Uncontrolled systemic illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-03; Primary Completion 2007-10 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Reduction in Young Mania Rating Scale score | Before and after intervention

SECONDARY OUTCOMES:
Clinical Global Impression | Before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Klein, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel